CLINICAL TRIAL: NCT03760081
Title: A Phase 2, Open-Label, Single-Arm, Multicenter Study to Assess the Safety and Efficacy of ASP1650, a Monoclonal Antibody Targeting Claudin 6 (CLDN6), in Male Subjects With Incurable Platinum Refractory Germ Cell Tumors
Brief Title: A Study to Assess the Safety and Efficacy of ASP1650, a Monoclonal Antibody Targeting Claudin 6 (CLDN6), in Male Subjects With Incurable Platinum Refractory Germ Cell Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1650-CL-0201
Record Dates: First submitted 2018-11-29; First posted 2018-11-30 (Actual); Results first posted 2021-11-10 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-10

CONDITIONS: Incurable Platinum Refractory Germ Cell Tumors; Tumors
Keywords: Incurable Platinum Refractory Germ Cell Tumors; ASP1650
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ASP1650, Dose Level 1 (Experimental): Participants received ASP1650 dose level 1 as intravenous infusion, every two weeks (Q2W) starting on Cycle 1 Day 1(C1D1) for up to a maximum of 12 cycles, or until disease progression, toxicity requiring study treatment cessation, start of another anticancer treatment, or until study discontinuation criteria was met, whichever occurred earlier. Duration of each treatment cycle was 14 days.
  Interventions: Drug: ASP1650
- ASP1650, Dose Level 2 (Experimental): Participants received ASP1650 dose level 2 as intravenous infusion, Q2W starting on C1D1 for up to a maximum of 12 cycles or until study discontinuation criteria as met, whichever occurred earlier. Duration of each treatment cycle was 14 days.
  Interventions: Drug: ASP1650

INTERVENTIONS:
Drug: ASP1650 — Participants received ASP1650 dose level 1 or dose level 2 as intravenous infusion, Q2W starting on C1D1 for up to a maximum of 12 cycles or until study discontinuation criterion was met, whichever occurred earlier. Duration of each treatment cycle was 14 days.

SUMMARY:
The purpose of this study was to establish the recommended phase 2 dose (RP2D) of ASP1650 (Safety Lead-in Phase), as well as, evaluate the efficacy of ASP1650 as measured by confirmed objective response rate (ORR) (phase 2) in participants with incurable platinum refractory germ cell tumors.

This study also evaluated the following efficacy measures for confirmed objective response rate (ORR); clinical benefit rate (CBR); duration of response (DOR); and progression-free survival (PFS); as well as safety and tolerability; the effect of ASP1650 on changes in serum beta human chorionic gonadotropin (βhCG) and alpha-fetoprotein (AFP); and the pharmacokinetics of ASP1650.

DETAILED DESCRIPTION:
The study consisted of 2 phases: Safety Lead-in phase and phase 2. 19 participants were enrolled in both phases.

The Safety Lead-in phase of this study was to establish the tolerability of RP2D. The RP2D determination was based on at least 6 evaluable participants at the RP2D as determined by the Dose Evaluation Committee (DEC).

Once RP2D had been established as tolerable, 13 additional participants were enrolled in phase 2 to receive ASP1650 for up to a maximum of 12 cycles or until a study discontinuation criteria had been met, whichever occurred earlier.

ELIGIBILITY:
Inclusion Criteria:

* A male subject with female partner(s) of child-bearing potential must agree to use contraception during the treatment period and for at least 6 months after the final study drug administration.
* Subject must not donate sperm during the treatment period and for 6 months after the final study treatment administration.
* A male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner is breastfeeding throughout the study period and for 6 months after the final study treatment administration.
* Subject agrees not to participate in another interventional study while receiving study drug in present study.

Disease Specific Criteria:

* Subject has histological evidence of germ cell tumor.
* Subject must have a germ cell tumor that is not amenable to cure with either surgery or chemotherapy.
* Subjects with seminoma and non-seminoma are eligible.
* Subject must have received initial cisplatin based combination chemotherapy AND demonstrated progression following at least 1 salvage regimen for advanced germ cell neoplasm (including relapsed primary mediastinal nonseminomatous germ cell tumor).

  1. Initial cisplatin based combination therapy includes bleomycin-etoposide-cisplatin, cisplatin-etoposide, etoposide-ifosfamide-cisplatin or similar regimens.
  2. "Salvage" regimens include high dose chemotherapy, paclitaxel-ifosfamide-cisplatin, vinblastine-ifosfamide cisplatin or similar regimens
  3. "Failure" of prior therapy is defined as: A > 25% increase in the products of perpendicular diameters of measurable tumor masses during prior therapy, which are not amenable to surgical resection; OR the presence of new tumor that are not amenable to surgical resection; OR an increase in alpha-fetoprotein (AFP) or beta human chorionic gonadotropin (βhCG) (≥ 50% increase in 2 separate samples collected at least 1 week apart are required if rising tumor markers are the only evidence of failure). NOTE: Subjects with clinically growing teratoma (enlarging mature teratoma arising during or after chemotherapy for a non seminomatous germ-cell tumor and with normal serum levels of AFP and βhCG) should undergo surgical resection if feasible.
* Subjects with late relapse (> 2 years) not amenable to resection are eligible.
* Subjects must have evidence of recurrent or metastatic carcinoma by 1 or more of the following:

  1. Subject has measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 within 28 days prior to the first dose of study treatment. For subjects with only 1 measurable lesion and prior radiotherapy, the lesion must be outside the field of prior radiotherapy or must have documented progression following radiation therapy.
  2. Subject has a baseline rising tumor marker (AFP or βhCG). NOTE: If a rising tumor marker is the only evidence of progressive disease, at least 2 consecutive rising values at least 1 week apart are needed. Subjects with only evidence of disease as rising tumor marker AFP and βhCG will be assessed for alternate causes of increased serum levels of these markers, such as cross reaction with luteinizing hormone (LH) (can be tested if needed by testosterone suppression of LH), hepatitis, use of marijuana or second primary tumor.

Physical or Laboratory Findings:

* Subject must have an available tumor specimen in a tissue block or unstained serial slides, or subject is an appropriate candidate for tumor biopsy and is amenable to undergoing a tumor biopsy during the screening period.
* Subject has Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Subject must meet all of the following criteria based on the centrally analyzed laboratory tests within 14 days prior to the first dose of study treatment. If repeat screening labs are required, local laboratory results can be used to confirm eligibility. In case of multiple central laboratory data within this period, the most recent data should be used to determine eligibility.

  1. Hemoglobin ≥ 8 g/dL
  2. Absolute neutrophil count (ANC) ≥ 1.0 x 109/L
  3. Platelets ≥ 75 x 109/L
  4. Albumin ≥ 2.5 g/dL
  5. Total bilirubin ≤ 2 x upper limit of normal (ULN) or direct bilirubin ≤ ULN for subjects with total bilirubin levels > 2 x ULN
  6. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN without liver metastases (or ≤ 5 x ULN if liver metastases are present)
  7. Estimated glomerular filtration rate ≥ 30 mL/min/1.73 m2
  8. Prothrombin time/international normalized ratio (PT/INR) and partial thromboplastin time (PTT) ≤ 2 x ULN (except for subjects receiving anticoagulation therapy)

Exclusion Criteria:

Prohibited Treatment or Therapies:

* Subject has received systemic immunosuppressive therapy, including systemic corticosteroids within 14 days prior to first dose of study treatment. Subject using a physiologic replacement dose of hydrocortisone or its equivalent (defined as up to 30 mg per day of hydrocortisone or up to 10 mg per day of prednisone) is eligible. Subject who received systemic steroids for asymptomatic central nervous system (CNS) metastases within 14 days prior to first dose of study treatment is eligible.
* Subject has received other investigational agents or devices within 28 days prior to first dose of study treatment.
* Subject has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., ≤ grade 1 or at baseline) from adverse event (AE) due to monoclonal antibody (mAb) agents administered more than 4 weeks earlier.
* Subject has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., ≤ grade 2 or at baseline) from AEs due to a previously administered agent.

Medical History or Concurrent Disease:

* Subject has prior severe allergic reaction or intolerance to a monoclonal antibody, including humanized or chimeric antibodies requiring permanent discontinuation.
* Subject has known immediate or delayed hypersensitivity, intolerance or contraindication to any component of study treatment.
* Subject has an active human immunodeficiency virus (HIV) infection or known active hepatitis B (HBsAg) or C infection. Subjects with well-controlled HIV infections (i.e., without detectable viral load) are eligible. For subjects who are negative for HBsAg, but hepatitis B core antibody (HBcAb) positive, an HBsAg deoxyribonucleic acid (DNA) test will be performed and if positive, the subject will be excluded. Subjects with positive serology but negative hepatitis C virus (HCV) ribonucleic acid (RNA) test results are eligible.
* Subject has active infection requiring systemic therapy that has not completely resolved within 14 days prior to first dose of study treatment.
* Subject has symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis. Subject with asymptomatic CNS metastases is eligible.
* Subject has had a major surgical procedure and has not completely recovered within 28 days prior to the first dose of study treatment.
* Subject has psychiatric illness or social situations that would preclude study compliance.
* Subject has another malignancy for which treatment is required. Subject with negligible risk of metastasis or death is eligible (e.g., basal or squamous cell skin cancer, localized prostate cancer treated with curative intent or incidental prostate cancer T1-T2a, Gleeson ≤ 3 + 4, PSA ≤ 0.5 and who are undergoing active surveillance).
* Subject has any concurrent disease, infection, or co-morbid condition that interferes with the ability of the subject to participate in the study, which places the subject at undue risk or complicates the interpretation of data.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (3):
- United States (3):
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Abramson Cancer Center University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Adra N, Vaughn DJ, Einhorn LH, Hanna NH, Funt SA, Rosales M, Arozullah A, Feldman DR. A phase II study assessing the safety and efficacy of ASP1650 in male patients with relapsed refractory germ cell tumors. Invest New Drugs. 2022 Oct;40(5):1087-1094. doi: 10.1007/s10637-022-01276-w. Epub 2022 Jun 27. PMID 35759134
- See also: Link to plain language summary of the study on the Trial Results Summaries website. — https://www.trialsummaries.com/Study/StudyDetails?id=14578&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 3 sites in the United States.
Pre-assignment Details: Adult male participants with incurable platinum refractory germ cell tumors for whom no standard of care treatment exists or who are ineligible to receive available standard of care treatment based on investigator's clinical judgment, who met all inclusion criteria and met none of the exclusion criteria were enrolled in this study. A total of 23 participants entered screening process and out of which 4 participants failed screened process.
Groups:
- ASP1650, Dose Level 1: Participants received ASP1650, dose level 1 as intravenous infusion, every two weeks (Q2W) starting on Cycle 1 Day 1 (C1D1) for up to a maximum of 12 cycles, or a until study discontinuation criteria was met, whichever occurred earlier. Duration of each treatment cycle was 14 days.
- ASP1650, Dose Level 2: Participants received ASP1650, dose level 2 as intravenous infusion, Q2W starting on C1D1 for up to a maximum of 12 cycles or until a study discontinuation criteria was met, whichever occurred earlier. Duration of each treatment cycle was 14 days.
Period: Overall Study
Arm/Group | ASP1650, Dose Level 1 | ASP1650, Dose Level 2
Started | 6 | 13
Completed | 0 | 1
Not Completed | 6 | 12
Not completed — Miscellaneous | 0 | 1
Not completed — Progressive Disease | 5 | 10
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF) population which included all enrolled participants who took at least 1 dose of ASP1650.
Groups:
- ASP1650, Dose Level 1: Participants received ASP1650, dose level 1 as intravenous infusion, Q2W starting on C1D1 for up to a maximum of 12 cycles, or until a study discontinuation criteria was met, whichever occurred earlier. Duration of each treatment cycle was 14 days.
- Total: Total of all reporting groups
Arm/Group | ASP1650, Dose Level 1 | ASP1650, Dose Level 2 | Total
Number analyzed (Participants) | 6 | 13 | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.8 (10.6) | 36.9 (12.2) | 37.2 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 13 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 5 | 10 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 13 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose (RP2D) of ASP1650
Description: The RP2D was determined via dose limiting toxicity (DLT) assessment by dose evaluation committee (DEC). DLT was evaluated according to National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTCAE) version 5.0.
Time Frame: Up to 28 days
Population: SAF population
Measure: Number; unit: Milligram per meter square (mg/m^2)
Groups:
- ASP1650: Participants received ASP1650, dose level 1 or dose level 2 as intravenous infusion, Q2W starting on C1D1 for up to a maximum of 12 cycles, or until a study discontinuation criteria was met, whichever occurred earlier. Duration of each treatment cycle was 14 days.
Arm/Group | ASP1650
Number analyzed (Participants) | 19
Milligram per meter square (mg/m^2) | 1500

2. Primary Outcome: Percentage of Participants With Confirmed Objective Response by Modified RECIST v1.1
Description: Confirmed objective response was defined as the confirmed completed response (CR) or confirmed partial response (PR), as confirmed by investigator based on modified Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Per modified RECIST v1.1, CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Both Alpha-Fetoprotein (AFP) and Beta Human Chorionic Gonadotropin (beta-HCG) values were below the ULN. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. No increase ≥ 50% in 2 samples at least 1 week apart compared to nadir values for both AFP and beta-HCG.
Time Frame: From randomization until confirmed CR or confirmed PR, whichever occurred first (up to 26.57 weeks)
Population: Full analysis set (FAS) population which included all enrolled participants.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | ASP1650, Dose Level 1 | ASP1650, Dose Level 2
Number analyzed (Participants) | 6 | 13
Percentage of participants | 0.0 [0.0 to 39.3] | 0.0 [0.0 to 20.6]

3. Secondary Outcome: Percentage of Participants With Confirmed Objective Response by RECIST v1.1
Description: Confirmed objective response was defined as the confirmed CR or PR, as confirmed by investigator based on RECIST v1.1. Per RECIST v1.1, CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From randomization until confirmed CR or confirmed PR, whichever occurred first (up to 26.57 weeks)
Population: FAS population
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | ASP1650, Dose Level 1 | ASP1650, Dose Level 2
Number analyzed (Participants) | 6 | 13
Percentage of participants | 0.0 [0.0 to 39.3] | 0.0 [0.0 to 20.6]

4. Secondary Outcome: Percentage of Participants With Clinical Benefit by Modified RECIST v1.1 and RECIST v1.1
Description: Clinical benefit: defined as best overall response of confirmed CR, confirmed PR, or durable stable disease (SD) as confirmed by investigator based on modified RECIST v1.1 and RECIST v1.1. Per RECIST v1.1 and modified RECIST V1.1, CR: disappearance of all target lesions. Any pathological lymph nodes(whether target or non-target) must have reduction in short axis to <10 mm. PR:at least a 30% decrease in sum of diameters of target lesions, taking as reference baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference smallest sum diameters while on study. Durable SD: SD maintained for at least 12 weeks. Additionally, per modified RECIST v1.1, CR also included AFP and beta-HCG values below ULN. PR also included no increase ≥ 50% in 2 samples at least 1 week apart compared to nadir values both for AFP and beta-HCG.
Time Frame: From randomization until confirmed CR, confirmed PR, or durable SD whichever occurred first (up to 26.57 weeks)
Population: FAS population
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | ASP1650, Dose Level 1 | ASP1650, Dose Level 2
Number analyzed (Participants) | 6 | 13
Percentage of participants
  Modified RECIST v1.1 | 0.0 [0.0 to 39.3] | 7.7 [0.4 to 31.6]
  RECIST v1.1 | 0.0 [0.0 to 39.3] | 7.7 [0.4 to 31.6]

5. Secondary Outcome: Duration of Response (DOR) by Modified RECIST v1.1 and RECIST v1.1 for Dose Level 2
Description: DOR was defined as the time from the date of the first confirmed response CR or confirmed PR (whichever was first recorded) as confirmed by investigator based on modified RECIST 1.1 and RECIST v1.1 to the date of disease progression or date of censoring, whichever was earlier. If a participant had not progressed, participant was censored at the date of last disease assessment or at the date of first confirmed CR/PR if no post-baseline disease assessment was available. DOR (in days) was calculated as: (Date of documented progressive disease [PD], death, or censoring) minus (Date of the first CR/PR which was subsequently confirmed) +1. Duration of response was planned to summarized only for participants receiving dose level 2 in phase 2.
Time Frame: From randomization until confirmed CR or confirmed PR whichever occurred first (up to 26.57 weeks)
Population: DOR was not analyzed since no participants had confirmed response of CR or PR in the study.
Arm/Group | ASP1650, Dose Level 2
Number analyzed (Participants) | 0

6. Secondary Outcome: Progression-Free Survival (PFS) by Modified RECIST v1.1 and RECIST v1.1 for Dose Level 2
Description: PFS was defined as the time from the date of first dose until the date of disease progression, or until death due to any cause. If a participant had neither progressed nor died, the participant was censored at the date of last disease as confirmed by investigator based on modified RECIST v1.1 and RECIST v1.1. The distribution of PFS was planned to be summarized only for participants receiving dose level 2 using Kaplan-Meier methodology. Per modified RECIST v1.1 and RECIST v1.1, Progressive disease (PD): appearance of one or more new lesions or at least a 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study (this includes the baseline sum if that is the smallest on study). Also, the sum must be an absolute increase of at least 5 mm. Additionally per modified RECIST v1.1, PD was increase ≥ 50% in serum tumor markers AFP or beta-hCG in 2 samples at least 1 week apart compared to nadir values.
Time Frame: From the date of first dose until the date of disease progression, or until death due to any cause (up to 26.57 weeks)
Population: FAS population
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | ASP1650, Dose Level 2
Number analyzed (Participants) | 13
Months
  Modified RECIST V1.1 | 1.18 [0.92 to 1.48]
  RECIST V1.1 | 1.45 [0.92 to 2.10]

7. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered with an Investigational Product (IP) which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign including abnormal laboratory finding/test result or other safety assessment, symptom, or disease temporally associated with use of IP whether or not considered related to IP. A treatment-emergent adverse event (TEAE) was defined as an AE with onset at any time from first dosing until last scheduled procedure. AEs were considered serious (SAEs) if AE resulted in death, was life-threatening, resulted in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, resulted in congenital anomaly, birth defect, or required inpatient hospitalization or led to prolongation of hospitalization.
Time Frame: From first dose of study drug up to 30 days after the last dose of study drug (up to 41.14 weeks)
Population: SAF population
Measure: Number; unit: Participants
Arm/Group | ASP1650, Dose Level 1 | ASP1650, Dose Level 2
Number analyzed (Participants) | 6 | 13
Participants
  TEAE | 5 | 13
  Drug-Related TEAEs | 2 | 5
  Serious TEAEs | 3 | 7
  Drug-Related Serious TEAE | 0 | 1
  TEAE Leading to Death | 1 | 3
  Drug-Related TEAE Leading to Death | 0 | 0
  TEAE Leading to Withdrawal of Treatment | 1 | 0
  Drug-Related TEAE Leading to Withdrawal of Treatment | 0 | 0
  Death | 3 | 5

8. Secondary Outcome: Number of Participants With Shifts From Baseline to Post Baseline in Eastern Cooperative Oncology Group Performance Status (ECOG PS)
Description: Number of participants with shifts from baseline to post baseline in ECOG PS levels were reported. ECOG has 6 levels (0-5). Level 0 is fully active, able to carry on all pre-disease performance without restriction; Level 1 is restricted in physically strenuous activity but ambulatory ad able to carry out work of a light or sedentary nature, e.g. light house work, office work; Level 2 is ambulatory and capable of all self care but unable to carry out any work activities; up and about more than 50% of waking hours; Level 3 is capable of only limited self care; confined to bed or chair more than 50% of waking hours; Level 4 is completely disabled; cannot carry on any self care; totally confined to bed or chair); and Level 5 is dead.
Time Frame: Baseline, C2D1, C3D1, C4D1, C5D1, C6D1, C7D1, C8D1, C9D1, C10D1, C11D1, C12D1 (Duration of each treatment cycle was 14 days)
Population: SAF population with available data at each time point.
Measure: Number; unit: Participants
Arm/Group | ASP1650, Dose Level 1 | ASP1650, Dose Level 2
Number analyzed (Participants) | 6 | 13
Participants
  ECOG PS : 0 (baseline) to 0 (C2D1): number analyzed (Participants) | 6 | 12
  ECOG PS : 0 (baseline) to 0 (C2D1) | 3 | 8
  ECOG PS : 0 (baseline) to 1 (C2D1): number analyzed (Participants) | 6 | 12
  ECOG PS : 0 (baseline) to 1 (C2D1) | 1 | 0
  ECOG PS : 1 (baseline) to 0 (C2D1): number analyzed (Participants) | 6 | 12
  ECOG PS : 1 (baseline) to 0 (C2D1) | 1 | 1
  ECOG PS : 1 (baseline) to 1 (C2D1): number analyzed (Participants) | 6 | 12
  ECOG PS : 1 (baseline) to 1 (C2D1) | 1 | 2
  ECOG PS : 2 (baseline) to 1 (C2D1): number analyzed (Participants) | 6 | 12
  ECOG PS : 2 (baseline) to 1 (C2D1) | 0 | 1
  ECOG PS : 0 (baseline) to 0 (C3D1): number analyzed (Participants) | 2 | 6
  ECOG PS : 0 (baseline) to 0 (C3D1) | 1 | 4
  ECOG PS : 0 (baseline) to 1 (C3D1): number analyzed (Participants) | 2 | 6
  ECOG PS : 0 (baseline) to 1 (C3D1) | 0 | 1
  ECOG PS : 1 (baseline) to 0 (C3D1): number analyzed (Participants) | 2 | 6
  ECOG PS : 1 (baseline) to 0 (C3D1) | 1 | 0
  ECOG PS : 1 (baseline) to 1 (C3D1): number analyzed (Participants) | 2 | 6
  ECOG PS : 1 (baseline) to 1 (C3D1) | 0 | 1
  ECOG PS : 0 (baseline) to 0 (C4D1): number analyzed (Participants) | 1 | 4
  ECOG PS : 0 (baseline) to 0 (C4D1) | 1 | 3
  ECOG PS : 1 (baseline) to 1 (C4D1): number analyzed (Participants) | 1 | 4
  ECOG PS : 1 (baseline) to 1 (C4D1) | 0 | 1
  ECOG PS : 0 (baseline) to 0 (C5D1): number analyzed (Participants) | 1 | 3
  ECOG PS : 0 (baseline) to 0 (C5D1) | 1 | 2
  ECOG PS : 1 (baseline) to 0 (C5D1): number analyzed (Participants) | 1 | 3
  ECOG PS : 1 (baseline) to 0 (C5D1) | 0 | 1
  ECOG PS : 0 (baseline) to 0 (C6D1): number analyzed (Participants) | 1 | 2
  ECOG PS : 0 (baseline) to 0 (C6D1) | 1 | 1
  ECOG PS : 1 (baseline) to 1 (C6D1): number analyzed (Participants) | 1 | 2
  ECOG PS : 1 (baseline) to 1 (C6D1) | 0 | 1
  ECOG PS : 0 (baseline) to 0 (C7D1): number analyzed (Participants) | 1 | 1
  ECOG PS : 0 (baseline) to 0 (C7D1) | 1 | 0
  ECOG PS : 1 (baseline) to 1 (C7D1): number analyzed (Participants) | 1 | 1
  ECOG PS : 1 (baseline) to 1 (C7D1) | 0 | 1
  ECOG PS : 0 (baseline) to 0 (C8D1): number analyzed (Participants) | 1 | 1
  ECOG PS : 0 (baseline) to 0 (C8D1) | 1 | 0
  ECOG PS : 1 (baseline) to 1 (C8D1): number analyzed (Participants) | 1 | 1
  ECOG PS : 1 (baseline) to 1 (C8D1) | 0 | 1
  ECOG PS : 0 (baseline) to 0 (C9D1): number analyzed (Participants) | 1 | 1
  ECOG PS : 0 (baseline) to 0 (C9D1) | 1 | 0
  ECOG PS : 1 (baseline) to 1 (C9D1): number analyzed (Participants) | 1 | 1
  ECOG PS : 1 (baseline) to 1 (C9D1) | 0 | 1
  ECOG PS : 1 (baseline) to 1 (C10D1): number analyzed (Participants) | 0 | 1
  ECOG PS : 1 (baseline) to 1 (C10D1) |  | 1
  ECOG PS : 1 (baseline) to 1 (C11D1): number analyzed (Participants) | 0 | 1
  ECOG PS : 1 (baseline) to 1 (C11D1) |  | 1
  ECOG PS : 1 (baseline) to 1 (C12D1): number analyzed (Participants) | 0 | 1
  ECOG PS : 1 (baseline) to 1 (C12D1) |  | 1

9. Secondary Outcome: Change From Baseline in Serum Beta Human Chorionic Gonadotropin (βhCG)
Description: Blood was drawn for the measurement of serum βhCG at day 1 of every cycle (14 day cycle) to align with imaging assessment until the participant develops radiological disease progression per RECIST v1.1 evaluation or starts other systemic anticancer treatment. To evaluate the effect of ASP1650 on changes in serum βhCG, disease response was derived for participants with elevated serum tumor markers at baseline using CR, PR and SD.
Time Frame: Baseline, Cycle 2 Day 1 (C2D1), C3D1, C4D1, C5D1, C6D1, C7D1, C8D1, C9D1, C10D1, C11D1, C12D1 (duration of each cycle was 14 days)
Population: FAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: International unit per liter (IU/L)
Arm/Group | ASP1650, Dose Level 1 | ASP1650, Dose Level 2
Number analyzed (Participants) | 6 | 13
International unit per liter (IU/L)
  Baseline | 32641.67 (70670.15) | 1198.00 (2293.97)
  Change at C2D1: number analyzed (Participants) | 6 | 12
  Change at C2D1 | 13847.50 (28555.07) | 2573.42 (4680.05)
  Change at C3D1: number analyzed (Participants) | 2 | 6
  Change at C3D1 | 105.50 (149.20) | -0.83 (2.04)
  Change at C4D1: number analyzed (Participants) | 1 | 4
  Change at C4D1 | 0.00 (NA) — Since only one participant was available for analysis at C4D1, standard deviation could not be calculated. | -1.25 (2.50)
  Change at C5D1: number analyzed (Participants) | 1 | 3
  Change at C5D1 | 0.00 (NA) — Since only one participant was available for analysis at C5D1, standard deviation could not be calculated. | -2.00 (3.46)
  Change at C6D1: number analyzed (Participants) | 1 | 2
  Change at C6D1 | 0.00 (NA) — Since only one participant was available for analysis at C6D1, standard deviation could not be calculated. | -1.00 (1.41)
  Change at C7D1: number analyzed (Participants) | 1 | 1
  Change at C7D1 | 0.00 (NA) — Since only one participant was available for analysis at C7D1, standard deviation could not be calculated. | 1.00 (NA) — Since only one participant was available for analysis at C7D1, standard deviation could not be calculated.
  Change at C8D1: number analyzed (Participants) | 1 | 1
  Change at C8D1 | 0.00 (NA) — Since only one participant was available for analysis at C8D1, standard deviation could not be calculated. | 2.00 (NA) — Since only one participant was available for analysis at C8D1, standard deviation could not be calculated.
  Change at C9D1: number analyzed (Participants) | 1 | 1
  Change at C9D1 | 0.00 (NA) — Since only one participant was available for analysis at C9D1, standard deviation could not be calculated. | 3.00 (NA) — Since only one participant was available for analysis at C9D1, standard deviation could not be calculated.
  Change at C10D1: number analyzed (Participants) | 0 | 1
  Change at C10D1 |  | -9.00 (NA) — Since only one participant was available for analysis at C10D1, standard deviation could not be calculated.
  Change at C11D1: number analyzed (Participants) | 0 | 1
  Change at C11D1 |  | 12.00 (NA) — Since only one participant was available for analysis at C11D1, standard deviation could not be calculated.
  Change at C12D1: number analyzed (Participants) | 0 | 1
  Change at C12D1 |  | 85.00 (NA) — Since only one participant was available for analysis at C12D1, standard deviation could not be calculated.

10. Secondary Outcome: Change From Baseline in Serum Alpha-Fetoprotein (AFP)
Description: Blood was drawn for the measurement of serum AFP at day 1 of every cycle (14 day cycle) to align with imaging assessment until the participant develops radiological disease progression per RECIST v1.1 evaluation or starts other systemic anticancer treatment. To evaluate the effect of ASP1650 on changes in serum AFP, disease response was derived for participants with elevated serum tumor markers at baseline using CR, PR and SD.
Time Frame: Baseline, C2D1, C3D1, C4D1, C5D1, C6D1, C7D1, C8D1, C9D1, C10D1, C11D1, C12D1 (duration of each cycle was 14 days)
Population: FAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: Microgram per liter (ug/L)
Arm/Group | ASP1650, Dose Level 1 | ASP1650, Dose Level 2
Number analyzed (Participants) | 6 | 13
Microgram per liter (ug/L)
  Baseline | 948.65 (2065.59) | 7116.52 (14580.47)
  Change at C2D1: number analyzed (Participants) | 6 | 12
  Change at C2D1 | -84.03 (257.70) | 2504.03 (6139.95)
  Change at C3D1: number analyzed (Participants) | 2 | 6
  Change at C3D1 | -8.00 (11.31) | 5404.50 (11064.94)
  Change at C4D1: number analyzed (Participants) | 1 | 4
  Change at C4D1 | 5.00 (NA) — Since only one participant was available for analysis at C4D1, standard deviation could not be calculated. | 2592.25 (4354.92)
  Change at C5D1: number analyzed (Participants) | 1 | 3
  Change at C5D1 | -8.00 (NA) — Since only one participant was available for analysis at C5D1, standard deviation could not be calculated. | 762.00 (1101.92)
  Change at C6D1: number analyzed (Participants) | 1 | 2
  Change at C6D1 | 99.00 (NA) — Since only one participant was available for analysis at C6D1, standard deviation could not be calculated. | 1343.00 (1650.39)
  Change at C7D1: number analyzed (Participants) | 1 | 1
  Change at C7D1 | 94.00 (NA) — Since only one participant was available for analysis at C7D1, standard deviation could not be calculated. | 118.00 (NA) — Since only one participant was available for analysis at C7D1, standard deviation could not be calculated.
  Change at C8D1: number analyzed (Participants) | 1 | 1
  Change at C8D1 | 138.00 (NA) — Since only one participant was available for analysis at C8D1, standard deviation could not be calculated. | 99.00 (NA) — Since only one participant was available for analysis at C8D1, standard deviation could not be calculated.
  Change at C9D1: number analyzed (Participants) | 1 | 1
  Change at C9D1 | 98.00 (NA) — Since only one participant was available for analysis at C9D1, standard deviation could not be calculated. | -27.00 (NA) — Since only one participant was available for analysis at C9D1, standard deviation could not be calculated.
  Change at C10D1: number analyzed (Participants) | 0 | 1
  Change at C10D1 |  | -454.00 (NA) — Since only one participant was available for analysis at C10D1, standard deviation could not be calculated.
  Change at C11D1: number analyzed (Participants) | 0 | 1
  Change at C11D1 |  | -579.10 (NA) — Since only one participant was available for analysis at C11D1, standard deviation could not be calculated.
  Change at C12D1: number analyzed (Participants) | 0 | 1
  Change at C12D1 |  | -598.90 (NA) — Since only one participant was available for analysis at C12D1, standard deviation could not be calculated.

11. Secondary Outcome: Pharmacokinetics (PK) of ASP1650 in Plasma: Area Under the Concentration-Time Curve Over 336 Hours (AUC336)
Description: AUC336 was derived from the Pharmacokinetic (PK) plasma samples collected. Duration of each cycle was 14 days.
Time Frame: Dose Level 1 - CID1, C3D1: predose, 1.5 h after start of infusion, immediately after end of infusion, 0.5, 1.5, 3, 6, 24, 48, 72 h after end of infusion; Dose Level 2 - C1D1, C3D1: predose, immediately after end of infusion
Population: Pharmacokinetic analysis set (PKAS) population with available data at each time point. PKAS population included all enrolled participants who took at least 1 dose of ASP1650 and for whom at least 1 ASP1650 concentration measurement was available.
Measure: Mean (Standard Deviation); unit: microgram*hour per milliliter (ug*h/mL)
Arm/Group | ASP1650, Dose Level 1 | ASP1650, Dose Level 2
Number analyzed (Participants) | 6 | 13
microgram*hour per milliliter (ug*h/mL)
  C1D1: number analyzed (Participants) | 5 | 10
  C1D1 | 73000 (25600) | 112000 (28300)
  C3D1: number analyzed (Participants) | 1 | 3
  C3D1 | 156000 (NA) — Since only one participant was available for analysis at C3D1, standard deviation could not be calculated. | 137000 (14800)

12. Secondary Outcome: Pharmacokinetics (PK) of ASP1650 in Plasma: Maximum Concentration (Cmax)
Description: Cmax was derived from the PK plasma samples collected. Duration of each cycle was 14 days.
Time Frame: Dose Level 1-CID1, C3D1: predose, 1.5 h after start of infusion, immediately after end of infusion, 0.5, 1.5, 3, 6, 24, 48, 72 h after end of infusion; Dose Level 2-C1D1, C3D1: predose, immediately after end of infusion
Population: PKAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (ug/mL)
Arm/Group | ASP1650, Dose Level 1 | ASP1650, Dose Level 2
Number analyzed (Participants) | 6 | 13
microgram per milliliter (ug/mL)
  C1D1 | 757 (245) | 1080 (277)
  C3D1: number analyzed (Participants) | 2 | 5
  C3D1 | 904 (NA) — Since very few participants were available for analysis at C3D1, standard deviation could not be calculated. | 1300 (227)

13. Secondary Outcome: Pharmacokinetics (PK) of ASP1650 in Plasma: Time to Maximum Concentration (Tmax)
Description: Tmax was derived from the PK plasma samples collected. Duration of each cycle was 14 days.
Time Frame: Dose Level 1- CID1, C3D1: predose, 1.5 h after start of infusion, immediately after end of infusion, 0.5, 1.5, 3, 6, 24, 48, 72 h after end of infusion; Dose Level 2- C1D1, C3D1: predose, immediately after end of infusion
Population: PKAS analysis with available data at each time point.
Measure: Median (Full Range); unit: hour
Arm/Group | ASP1650, Dose Level 1 | ASP1650, Dose Level 2
Number analyzed (Participants) | 6 | 13
hour
  C1D1 | 2.03 [2.00 to 2.50] | 4.50 [3.08 to 9.00]
  C3D1: number analyzed (Participants) | 2 | 5
  C3D1 | 3.38 [2.00 to 4.75] | 3.50 [3.05 to 4.50]

14. Secondary Outcome: Pharmacokinetics (PK) of ASP1650 in Plasma: Concentration Immediately Prior to Dosing at Multiple Dosing (Ctrough)
Description: Ctrough was derived from the PK plasma samples collected. Duration of each cycle was 14 days.
Time Frame: C2D1,C3D1,C4D1,C5D1,C6D1,C7D1,C8D1,C9D1,C10D1,C11D1,C12D1:predose,1.5 h post start of infusion, immediately post end of infusion,0.5,1.5,3,6,24,48,72 h post end of infusion for Dose Level 1, and predose, immediately post end of infusion for Dose Level 2
Population: PKAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | ASP1650, Dose Level 1 | ASP1650, Dose Level 2
Number analyzed (Participants) | 6 | 13
ug/mL
  C2D1: number analyzed (Participants) | 6 | 11
  C2D1 | 74.55 (62.79) | 111.64 (44.59)
  C3D1: number analyzed (Participants) | 1 | 5
  C3D1 | 238 (NA) — Since only one participant was available for analysis at C3D1, standard deviation could not be calculated. | 163.6 (39.16)
  C4D1: number analyzed (Participants) | 1 | 4
  C4D1 | 290 (NA) — Since only one participant was available for analysis at C4D1, standard deviation could not be calculated. | 184.5 (56.7)
  C5D1: number analyzed (Participants) | 1 | 3
  C5D1 | 343 (NA) — Since only one participant was available for analysis at C5D1, standard deviation could not be calculated. | 186.33 (39.55)
  C6D1: number analyzed (Participants) | 1 | 2
  C6D1 | 306 (NA) — Since only one participant was available for analysis at C6D1, standard deviation could not be calculated. | 232.5 (20.51)
  C7D1: number analyzed (Participants) | 1 | 1
  C7D1 | 317 (NA) — Since only one participant was available for analysis at C7D1, standard deviation could not be calculated. | 225 (NA) — Since only one participant was available for analysis at C7D1, standard deviation could not be calculated.
  C8D1: number analyzed (Participants) | 1 | 1
  C8D1 | 329 (NA) — Since only one participant was available for analysis at C8D1, standard deviation could not be calculated. | 200 (NA) — Since only one participant was available for analysis at C8D1, standard deviation could not be calculated.
  C9D1: number analyzed (Participants) | 1 | 1
  C9D1 | 318 (NA) — Since only one participant was available for analysis at C9D1, standard deviation could not be calculated. | 296 (NA) — Since only one participant was available for analysis at C9D1, standard deviation could not be calculated.
  C10D1: number analyzed (Participants) | 0 | 1
  C10D1 |  | 223 (NA) — Since only one participant was available for analysis at C10D1, standard deviation could not be calculated.
  C11D1: number analyzed (Participants) | 0 | 1
  C11D1 |  | 21.3 (NA) — Since only one participant was available for analysis at C11D1, standard deviation could not be calculated.
  C12D1: number analyzed (Participants) | 0 | 1
  C12D1 |  | 82.4 (NA) — Since only one participant was available for analysis at C12D1, standard deviation could not be calculated.

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after the last dose of study drug (up to 41.14 weeks)
Arm/Group | ASP1650, Dose Level 1 | ASP1650, Dose Level 2
All-Cause Mortality (participants affected / at risk) | 3/6 | 5/13
Serious Adverse Events (participants affected / at risk) | 3/6 | 7/13
Other Adverse Events (participants affected / at risk) | 5/6 | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | ASP1650, Dose Level 1 (N=6) | ASP1650, Dose Level 2 (N=13)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0/6 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Abdominal infection (Infections and infestations) | 0 (0) | 1/6 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 1/6 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0/6 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | ASP1650, Dose Level 1 (N=6) | ASP1650, Dose Level 2 (N=13)
Anaemia (Blood and lymphatic system disorders) | 3 (7) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1/6 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1/6 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1/6 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1/6 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0/6 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0/6 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1/6 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1/6 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0/6 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0/6 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1/6 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0/6 (0)
Hypertension (Vascular disorders) | 1 (4) | 0/6 (0)
Hypotension (Vascular disorders) | 0 (0) | 1/6 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
Blood testosterone decreased (Investigations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Oedema genital (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2020-04-17): https://cdn.clinicaltrials.gov/large-docs/81/NCT03760081/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT03760081/SAP_001.pdf